CLINICAL TRIAL: NCT00639288
Title: Modification of Cognitive Processing Therapy (CPT-C) for Posttraumatic Stress Disorder (PTSD) and Alcohol Dependence (AD)
Brief Title: Modification of Cognitive Processing Therapy (CPT-C) for PTSD and Alcohol Dependence
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IP0036; MIRECC
Record Dates: First submitted 2008-03-13; First posted 2008-03-20 (Estimated); Last update posted 2016-03-21 (Estimated); Status verified 2016-03

CONDITIONS: Alcohol Dependence; PTSD
Keywords: Alcohol Dependence; PTSD; CPT-C
MeSH Terms: conditions — Alcoholism; Stress Disorders, Post-Traumatic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): modified CPT-C
  Interventions: Other: modified CPT-C

INTERVENTIONS:
Other: modified CPT-C — modified CPT-C

SUMMARY:
Objective: To develop a detailed treatment manual that modifies the existing CPT-C treatment protocol to allow for concurrent treatment of PTSD and AD, and to obtain some pilot data regarding its efficacy.

Hypothesis: We predict that CPT-C will significantly reduce the number of drinking days (measured by the Timeline Follow Back Method [TLFB]) and reduce the symptoms of PTSD (measured by the [CAPS and PCL] scores).

Design: This is a non-randomized, prospective study in which all participants will receive the modified CPT-C for 12 weeks by trained CPT-C clinicians, with each session lasting approximately 1-1.5 hours). Modifications to CPT-C include psychoeducation about alcohol use as an avoidance of PTSD symptoms integrated throughout treatment, integration of coping skills training for AD, weekly breathalyzer tests to measure blood alcohol level, and use and collection of daily dairies of alcohol use.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females between the ages of 21-65 years old.
2. Current alcohol dependence as determined by the Structured Clinical Interview for DSM-IV Axis I Disorder (SCID; First et al. 1996). Abstinence no more than past 29 days. Primary substance dependence diagnosis of alcohol dependence.
3. Current PTSD as determined by the Clinician Administered PTSD Scale for DSM-IV(CAPS; Blake et al. 1995).
4. Participants on psychiatric medication must be on a stable regimen for at least 2 weeks before treatment begins.
5. Ability to participate psychologically and physically, able to give informed consent and complete assessments, and participate in study procedures.

Exclusion Criteria:

1. Current psychotic disorders
2. Current suicidal or homicidal ideations
3. Current substance dependence other than alcohol or nicotine dependence
4. Legal charges pending with potential of incarceration
5. Unstable serious medical conditions or one requiring acute medical treatments or anticipation of hospitalization for extended care

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2008-03; Primary Completion 2014-10 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Alcohol use, PTSD symptoms | 16 weeks

SECONDARY OUTCOMES:
quality of life | 16 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Ismene L Petrakis, MD, Principal Investigator — Yale University
Locations (1):
- VA Connecticut Healthcare System - West Haven Campus, West Haven, Connecticut, United States